CLINICAL TRIAL: NCT03330652
Title: Identifying Health Disparities and Health Services Gaps by Following Stroke Patients and Their Family Care-givers to Explore Their Needs and Expectations: A Multi-center Longitudinal Study
Brief Title: Health Disparities in Stroke Patients and Their Families: a Longitudinal Multicenter Study (HDSS)
Acronym: HDSS
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Israel National Institute for Health Policy and Health Services Research (Other Government)
Responsible Party: Principal Investigator, Dr. Rachel Dankner, Principal Investigator, Sheba Medical Center
Other Study IDs: SHEBA-16-2912-RD-CTIL
Record Dates: First submitted 2017-10-15; First posted 2017-11-06 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2020-08

CONDITIONS: Stroke, Acute
Keywords: Quality of life; Cognitive function; Mental state; Functional capacity; EQ5D; HADS; Barthel Index; mRS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The meeting point of the patient and his/her immediate family with the health care system is complicated and traumatic. While having to deal with medicalization geared towards providing evidence-based and cost-effective medical care, the patient expects comprehensive, holistic care tailored to his/her needs, during hospitalization or in the community. A survey of 800 stroke patients and their caregiver during the 1st year following acute stroke hospitalization will explore their unmet needs.

DETAILED DESCRIPTION:
Background: The meeting point of the patient with the health care system is complicated and traumatic. The patient's autonomy over physical health becomes diminished. The patient and his family need to deal with medicalization geared towards providing evidence-based medical care, while attempting to be cost-efficient. The patient expects comprehensive, holistic care tailored to his/her needs, during hospitalization or in the community.

Objectives: To characterize the patient's and his/her family's needs and expectations from the medical system, following an acute medical event involving hospitalization and community care treatment; to analyze the gaps between these needs and the actual treatment provided.

Working hypotheses: Certain needs and expectations of patients and their families are unrecognized and unmet by the medical system; more deprived population groups can be identified, where the gap between needs and service provided is exceptionally great.

Type of research and methods of data collection: Prospective cohort study. Method(s) of data collection: 800 stroke patients hospitalized at 4 medical centers: Tel Hashomer, Soroka, Asaf-Harofeh, and Naharia, and a close family member (caregiver), will be recruited during one calendar year. These medical centers reflect the heterogeneity of the population, it's ethnic diversity, and the periphery vs. the central areas of the country of Israel. Personal details will be recorded, and informed consent forms signed. The patients will be telephone-interviewed 3-4 months after acute hospitalization, 6-8 months, and after one year, to assess their functionality, coping with bureaucracy, availability and accessibility (financial and cultural), disease management, continuity of treatment, number of caregivers, quality of life, depression, cognitive function, care received by the medical system, "patient at the center" assessment.

Uniqueness and relevance to the National health Insurance Law: Assessment of patient's experience (and his caregivers) in the first year after hospitalization due to stroke, with emphasis on inequality between patients based on socio-economic factors. The assumption is that the gap between expectations and needs of patient and family from the medical system and actual service provided by the system is even bigger among populations who depend more on the system for support.

Among the Ministry of Health's 6 pillars of health is reinforcement of the perception of "patient-centered care" which aims to map out gaps, reasons and challenges in putting this objective into practice. Findings of this research will enable decision makers to efficiently allocate resources and funds to needy populations, thus reducing gaps, lowering use of the medical system and lowering costs incurred by the system.

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke
* Caregiver of patient who's an immediate family member

Exclusion Criteria:

* Inability to communicate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 800 stroke patients/spouces hospitalized at 4 medical centers, and a close family member, will be recruited during one calendar year.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
"patient at the center" assessment | 12 months after acute stroke
  coping with bureaucracy, availability and accessibility (financial and cultural), disease management, continuity of treatment

SECONDARY OUTCOMES:
Change over the year of follow up in quality of life | 4, 8, 12 months after acute stroke
  Quality of life will be measured using the European Quality of life 5 Dimention (EQ5D) questionnaire. Scores range from 0-15 where 15 is the worst score
Change over the year of follow up in mental health | 4, 8, 12 months after acute stroke
  Mental health will be evaluated for anxiety and depression using the Hospital and Anxiety Disease Scale (HADS). Score range 0-21 for each anxiety and depression subscales. 21 means worst score.
Change over the year of follow up in functional capacity | 4, 8, 12 months after acute stroke
  Functional capacity of the stroke patient will be measured using the Barthel index. Scores range 0-100 where 0 means worst dissability.
Change over the year of follow up in burden of care | 4, 8, 12 months after acute stroke
  Burden of care as it is experienced by the caregiver of the stroke patient will be evaluated by the Zarit questionnaire. A scale of 0-88 where 88 means the most severe burden

CONTACTS AND LOCATIONS:
Overall Officials: Rachel S Dankner, MD, MPH, Principal Investigator — The Gertner Institute
Locations (4):
- Israel (4):
  - Neurologic Department, Barzilai Medical Center, Ashkelon
  - Neurologic Department, Soroka Medical Center, Beersheba
  - Neurologic Department, El Hagalil Medical Center, Nahariya
  - Neurologic Department, Sheba Medical Center, Ramat Gan